CLINICAL TRIAL: NCT07111078
Title: VRC 329: A Phase I Open-Label, Clinical Trial to Evaluate the Safety, Tolerability, and Immunogenicity of a Quadrivalent Influenza HA Stem Vaccine VRC-FLUMOS0122-00-VP (STEMos1) With and Without ALFQ Adjuvant in Healthy Adults
Brief Title: Quadrivalent Influenza HA Stem Vaccine VRC-FLUMOS0122-00-VP (SteMos1) With and Without ALFQ Adjuvant in Healthy Adults
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Prevention
Other Study IDs: 10002425; 002425-I
Record Dates: First submitted 2025-08-07; First posted 2025-08-08 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01-16

CONDITIONS: Influenza Prevention; Pandemic Influenza Prevention
Keywords: Dose-Escalation; INFLUENZA VIRUS; Immune Response; Respiratory Illness; Experimental Vaccine; Safety
MeSH Terms: interventions — Adjuvants, Pharmaceutic

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Group 1 (Experimental): 60 mcg of SteMos1 on Day 0 and Week 16
  Interventions: Biological: VRC-FLUMOS0122-00-VP (SteMos1) with and without Army Liposome Formulation containing saponin QS-21 (ALFQ) Adjuvant
- Group 2 (Experimental): 180 mcg of SteMos1 on Day 0 and Week 16
  Interventions: Biological: VRC-FLUMOS0122-00-VP (SteMos1) with and without Army Liposome Formulation containing saponin QS-21 (ALFQ) Adjuvant
- Group 3 (Experimental): 60 mcg of SteMos1 + 0.5 ml of ALFQ on Day 0 and Week 16
  Interventions: Biological: VRC-FLUMOS0122-00-VP (SteMos1) with and without Army Liposome Formulation containing saponin QS-21 (ALFQ) Adjuvant
- Group 4 (Experimental): 180 mcg of SteMos1 + 0.5 ml of ALFQ on Day 0 and Week 16
  Interventions: Biological: VRC-FLUMOS0122-00-VP (SteMos1) with and without Army Liposome Formulation containing saponin QS-21 (ALFQ) Adjuvant
- Group 5- optional (Experimental): SteMos1 [dose TBD based on interim analysis of data from Groups 3-4] + 0.5 ml of ALFQ on Day 0 and Week 16
  Interventions: Biological: VRC-FLUMOS0122-00-VP (SteMos1) with and without Army Liposome Formulation containing saponin QS-21 (ALFQ) Adjuvant

INTERVENTIONS:
Biological: VRC-FLUMOS0122-00-VP (SteMos1) with and without Army Liposome Formulation containing saponin QS-21 (ALFQ) Adjuvant — FLUMOS0122-00-VP (SteMos1) is a sterile, aqueous buffered solution supplied in 3 mL single-dose glass vials containing 0.7 +/- 0.1 mL with a vaccine concentration of 1080 mcg/mL.
  The ALFQ drug product is a sterile suspension that contains 240 mcg of monophosphoryl 3-deacyl Lipid A (3D-PHAD) and 120 mcg QS-21 that is vialed at 0.6 mL/vial in 3.0 mL glass vials. 0.5 mL of ALFQ adjuvant will be mixed with the 60 or 180 mcg dose of SteMos1 during preparation in the pharmacy prior to

SUMMARY:
Background:

Influenza (flu) is a contagious respiratory illness caused by viruses. Flu symptoms can range from mild to severe, and the illness can be fatal. Vaccines help the body learn to prevent or fight infections such as flu. Some vaccines are combined with adjuvants. Adjuvants are special salts or fats that help vaccines work better. Researchers are looking for ways to make flu vaccines more effective.

Objective:

To test a new flu vaccine with and without a new adjuvant.

Eligibility:

Healthy adults aged 18 to 50. They must have had at least 1 flu vaccine since 2020.

Design:

Participants will have 12 clinic visits over 15 months.

The vaccine is given as an injection into the muscle of the upper arm. Participants will be vaccinated during 2 visits spaced 4 months apart. Half will receive just the vaccine; half will receive the vaccine plus the adjuvant. They will be monitored for at least 30 minutes after each shot.

Participants will keep a diary for 7 days after each shot. They check their temperature every day and record any symptoms.

Participants will have 10 follow-up clinic visits plus 4 phone calls. They will have 4 to 10 tablespoons of blood drawn at each clinic visit. Fluid samples will be collected from their nose and mouth. They will be checked for any health changes.

Participants may opt to undergo apheresis: Blood will be taken from the body through a needle inserted into a vein. The blood will pass through a machine that separates out the white blood cells. The remaining blood will be returned to the body through a different needle.

DETAILED DESCRIPTION:
Design:

This is a phase I, open-label, dose escalation study to evaluate the safety, tolerability, and immunogenicity of the stem quadrivalent influenza vaccine VRC-FLUMOS0122-00-VP (SteMos1) with and without Army Liposome Formulation containing saponin QS-21 (ALFQ) adjuvant. The hypotheses are that the SteMos1 vaccine is safe and tolerable when administered alone or with ALFQ adjuvant, that this vaccine elicits vaccine specific immune responses, and that addition of the ALFQ adjuvant increases the magnitude and breadth of the elicited immune responses. The primary objective is to evaluate the safety and tolerability of the investigational vaccine with and without ALFQ adjuvant in healthy adults. Secondary objectives are related to the immunogenicity of the investigational vaccine with and without ALFQ adjuvant.

Study Products:

The investigational vaccine, SteMos1, was developed by the Vaccine Research Center (VRC), National Institute of Allergy and Infectious Diseases (NIAID). The adjuvant, Army Liposome Formulation containing QS-21 (ALFQ), was developed and provided by the Walter Reed Army Institute of Research (WRAIR).

The SteMos1 vaccine includes stabilized HA stems from the following 4 influenza strains:

Influenza A:

Group 1:

H2: A/Singapore/1/1957

H5: A/lndonesia/5/2005

Group 2:

H7: A/Anhui/1/2013

H10: A/Jiangxi-Donghu/346/2013

Participants:

Healthy adults 18-50 years of age, inclusive, will be enrolled

Study Plan:

There will be multiple interim safety reviews in this trial. The first review will assess the safety data for Group 1 (60 mcg of SteMos1 alone). Enrollment for Group 1 will be limited to one participant per day for the first three participants. After the third participant's two-week post-vaccination visit, a safety review will determine whether to continue enrollment at the same dose level in Group 1 and to proceed with enrollment of the next dose level, Group 2 (180 mcg of SteMos1 alone), and Group 3 (60 mcg of SteMos1 with ALFQ adjuvant). Group 2 and Group 3 will also enroll one participant per day for the first three participants in each group. Following the two-week post-vaccination visit of the third participant in each group, a safety review will determine whether to continue enrollment at the same dose level in Group 2 and Group 3 and to proceed to the next dose level, Group 4 (180 mcg of SteMos1 with ALFQ adjuvant). At this stage, these interim safety reviews for Group 2 and Group 3 can be conducted simultaneously or at different times, depending on which group first completes enrollment of the initial three participants.

Group 4 will enroll one participant per day for the first three participants. After the two-week post-vaccination visit of the third participant, a final safety review will determine whether to continue enrollment at the same dose level in Group 4. The study will not enroll any participants in Group 5 until available interim safety data from Group 3 and Group 4 are evaluated to select the dose for Group 5.

Once all groups are open, participants will be enrolled at the discretion of the Principal Investigator (PI) to balance enrollments in each group. If a current participant is discontinued from the protocol, a new participant may be enrolled at the discretion of the PI to collect required safety or immunogenicity data.

Solicited reactogenicity will be evaluated using a 7-day diary card. Assessment of vaccine safety will include clinical observation and monitoring of hematological and chemical parameters at clinical visits throughout the study.

Study Duration:

Participants will be followed for safety for a total time of 68 weeks, including through the 2025-2026 influenza season. This safety follow-up includes 52 weeks after the second dose of vaccine.

ELIGIBILITY:
* INCLUSION CRITERIA:

A participant must meet all of the following criteria:

* Healthy adults between the ages of 18-50 years, inclusive
* Based on history and physical examination, be in good general health and without a history of any of the conditions listed in the exclusion criteria
* Received at least one licensed influenza vaccine from the 2020-2021 influenza season through the 2024-2025 influenza season
* Able and willing to complete the informed consent process
* The ability to read and comprehend English as all consent and recruitment materials are in English.
* Available for clinic visits for 68 weeks after the first dose, including through the 2025-2026 influenza season
* Able to provide proof of identity to the satisfaction of the study clinician completing the enrollment process
* Physical examination and laboratory results without clinically significant findings and a Body Mass Index (BMI) <= 35 within the 56 days before enrollment
* Agrees to not receive any licensed influenza vaccination during study participation due to potential confounding of study results
* Willing to have blood and mucosal samples collected, stored indefinitely, and used for research purposes.

Laboratory Criteria within 56 days before enrollment:

* WBC and differential within institutional normal range or accompanied by approval of the site Principal Investigator (PI) or designee
* Total lymphocyte count >= 800 cells/microliter
* Platelets = 125,000-400,000 cells/mircoliter
* Hemoglobin within institutional normal range or accompanied by approval of the PI or designee
* Alanine aminotransferase (ALT) <= 1.25 x institutional upper limit of normal (ULN)
* Aspartate aminotransferase (AST) <= 1.25 x institutional ULN
* Alkaline phosphatase (ALP) < 1.1 x institutional ULN
* Total bilirubin within institutional normal range or accompanied by approval of the PI or designee
* Serum creatinine <= 1.1 x institutional ULN
* Negative for HIV infection by an FDA-approved method of detection

Criteria applicable to women of childbearing potential:

* Negative beta-human chorionic gonadotropin (beta-HCG) pregnancy test (urine or serum) on the day of enrollment
* Agrees to use an effective means of birth control from at least 21 days prior to enrollment through the end of the study

EXCLUSION CRITERIA:

Participant will be excluded if one or more of the following conditions apply:

-Women who are breast-feeding or planning to become pregnant during the study

A participant has received any of the following substances:

* Receipt of any licensed influenza vaccine or lab-confirmed influenza infection within 6 months prior to enrollment.
* Plan to or are required to receive the 2025-2026 or 2026-2027 licensed influenza vaccines
* Live attenuated vaccines within 4 weeks prior to enrollment
* Inactivated vaccines within 2 weeks prior to enrollment
* mRNA vaccines within 4 weeks prior to enrollment
* Receipt of the HA ferritin influenza vaccine VRC-FLUNPF081-00-VP alone or in prime-boost regimens with VRC-FLUDNA082-00-VP (HA-F A/Sing, DNA A/Sing, VRC 316).
* Receipt of the mosaic quadrivalent influenza vaccine VRC-FLUMOS0111-00-VP (FluMos-v1, VRC 325)
* Receipt of the mosaic hexavalent influenza vaccine VRC-FLUMOS0116-00-VP (FluMos-v2, VRC 326)
* More than 10 days of systemic immunosuppressive medications or cytotoxic medications within the 4 weeks prior to enrollment or any within the 14 days prior to enrollment
* Blood products within 16 weeks prior to enrollment
* Investigational research agents within 4 weeks prior to enrollment or planning to receive investigational products while on the study
* Current allergy treatment with allergen immunotherapy with antigen injections, unless on maintenance schedule
* Current anti-TB prophylaxis or therapy

Participant has a history of any of the following clinically significant conditions:

* Serious reactions to vaccines that preclude receipt of the study vaccinations as determined by the PI or designee
* Hereditary angioedema, acquired angioedema, or idiopathic forms of angioedema
* Asthma that is not well controlled
* Diabetes mellitus (type I or II), except for gestational diabetes
* Thyroid disease that is not well controlled
* Idiopathic urticaria within the past year
* Immune-mediated diseases, such as autoimmune or autoinflammatory diseases, or immunodeficiencies
* Hypertension that is not well controlled
* Bleeding disorder diagnosed by a doctor (e.g., factor deficiency, coagulopathy, or platelet disorder requiring special precautions) or significant bruising or bleeding difficulties with IM injections or blood draws
* Malignancy that is active or history of malignancy that is likely to recur during the period of the study
* Seizure disorder other than 1) febrile seizures, 2) seizures secondary to alcohol withdrawal more than 3 years ago, or 3) seizures that have not required treatment within the last 3 years
* Asplenia, functional asplenia or any condition resulting in the absence or removal of the spleen
* Guillain-Barr(SqrRoot)(Copyright) Syndrome
* Any medical, social condition, occupational reason, or other reason that, in the judgment of the PI or designee, is a contraindication to protocol participation or impairs a participant's ability to give informed consent, including but not limited to clinically significant forms of infectious diseases, drug or alcohol abuse, autoimmune diseases, psychiatric disorders, or heart disease.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 56 (Estimated)
Dates: Start 2025-08-27 (Actual); Primary Completion 2027-08-18 (Estimated); Study Completion 2027-08-18 (Estimated)

PRIMARY OUTCOMES:
To evaluate the safety and tolerability of SteMos1 (60 mcg) vaccine without ALFQ adjuvant administered as a 2-dose regimen | Though 52 weeks after the second vaccine administration
  Solicited reactogenicity will be evaluated using a 7-day diary card. Assessment of vaccine safety will include clinical observation and monitoring of hematological and chemical parameters at clinical visits throughout the study.
To evaluate the safety and tolerability of SteMos1 (180 mcg) vaccine without ALFQ adjuvant administered as a 2-dose regimen | Though 52 weeks after the second vaccine administration
  Solicited reactogenicity will be evaluated using a 7-day diary card. Assessment of vaccine safety will include clinical observation and monitoring of hematological and chemical parameters at clinical visits throughout the study.
To evaluate the safety and tolerability of SteMos1 (60 mcg) vaccine with ALFQ adjuvant administered as a 2-dose regimen | Though 52 weeks after the second vaccine administration
  Solicited reactogenicity will be evaluated using a 7-day diary card. Assessment of vaccine safety will include clinical observation and monitoring of hematological and chemical parameters at clinical visits throughout the study.
To evaluate the safety and tolerability of SteMos1 (180 mcg) vaccine with ALFQ adjuvant administered as a 2-dose regimen | Though 52 weeks after the second vaccine administration
  Solicited reactogenicity will be evaluated using a 7-day diary card. Assessment of vaccine safety will include clinical observation and monitoring of hematological and chemical parameters at clinical visits throughout the study.

SECONDARY OUTCOMES:
Antibody responses to SteMos1 (180 mcg) vaccine administered without ALFQ as a 2-dose regimen | Two weeks after each injection
  Binding antibody responses
Antibody responses to SteMos1 (60 mcg) vaccine administered without ALFQ as a 2-dose regimen | Two weeks after each injection
  Binding antibody responses
Antibody responses to SteMos1 (60 mcg) vaccine administered with ALFQ as a 2-dose regimen | Two weeks after each injection
  Binding antibody responses
Antibody responses to SteMos1 (180 mcg) vaccine administered with ALFQ as a 2-dose regimen | Two weeks after each injection
  Binding antibody responses

CONTACTS AND LOCATIONS:
Overall Officials: Lesia K Dropulic, M.D., Principal Investigator — National Institute of Allergy and Infectious Diseases (NIAID)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ober Shepherd BL, Scott PT, Hutter JN, Lee C, McCauley MD, Guzman I, Bryant C, McGuire S, Kennedy J, Chen WH, Hajduczki A, Mdluli T, Valencia-Ruiz A, Amare MF, Matyas GR, Rao M, Rolland M, Mascola JR, De Rosa SC, McElrath MJ, Montefiori DC, Serebryannyy L, McDermott AB, Peel SA, Collins ND, Joyce MG, Robb ML, Michael NL, Vasan S, Modjarrad K; EID-030 Study Group. SARS-CoV-2 recombinant spike ferritin nanoparticle vaccine adjuvanted with Army Liposome Formulation containing monophosphoryl lipid A and QS-21: a phase 1, randomised, double-blind, placebo-controlled, first-in-human clinical trial. Lancet Microbe. 2024 Jun;5(6):e581-e593. doi: 10.1016/S2666-5247(23)00410-X. Epub 2024 May 15. PMID 38761816
- [Background] Boyoglu-Barnum S, Ellis D, Gillespie RA, Hutchinson GB, Park YJ, Moin SM, Acton OJ, Ravichandran R, Murphy M, Pettie D, Matheson N, Carter L, Creanga A, Watson MJ, Kephart S, Ataca S, Vaile JR, Ueda G, Crank MC, Stewart L, Lee KK, Guttman M, Baker D, Mascola JR, Veesler D, Graham BS, King NP, Kanekiyo M. Quadrivalent influenza nanoparticle vaccines induce broad protection. Nature. 2021 Apr;592(7855):623-628. doi: 10.1038/s41586-021-03365-x. Epub 2021 Mar 24. PMID 33762730
- [Background] Widge AT, Hofstetter AR, Houser KV, Awan SF, Chen GL, Burgos Florez MC, Berkowitz NM, Mendoza F, Hendel CS, Holman LA, Gordon IJ, Apte P, Liang CJ, Gaudinski MR, Coates EE, Strom L, Wycuff D, Vazquez S, Stein JA, Gall JG, Adams WC, Carlton K, Gillespie RA, Creanga A, Crank MC, Andrews SF, Castro M, Serebryannyy LA, Narpala SR, Hatcher C, Lin BC, O'Connell S, Freyn AW, Rosado VC, Nachbagauer R, Palese P, Kanekiyo M, McDermott AB, Koup RA, Dropulic LK, Graham BS, Mascola JR, Ledgerwood JE; VRC 321 study team. An influenza hemagglutinin stem nanoparticle vaccine induces cross-group 1 neutralizing antibodies in healthy adults. Sci Transl Med. 2023 Apr 19;15(692):eade4790. doi: 10.1126/scitranslmed.ade4790. Epub 2023 Apr 19. PMID 37075129
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_002425-I.html